CLINICAL TRIAL: NCT02320214
Title: A Single-Center, Clinical Study to Evaluate the Safety of a Fragranced Personal Lubricant in Healthy Female Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Church & Dwight Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ST-7555
Record Dates: First submitted 2014-12-09; First posted 2014-12-19 (Estimated); Results first posted 2016-09-20 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-10

CONDITIONS: Erythema; Edema
MeSH Terms: conditions — Erythema; Edema

ARMS (1):
- Miami w/ frag Personal lubricant (Experimental): Healthy subjects use Novel lubricant Miami w/ frag Personal lubricant at least 4 times per week for 2 weeks.
  Interventions: Device: Miami w/ frag Personal lubricant

INTERVENTIONS:
Device: Miami w/ frag Personal lubricant

SUMMARY:
To evaluate the safety of Miami w/ frag Personal lubricant when used as indicated as a personal lubricant in the vagina and vulvar/perineal areas at least four times weekly for two weeks in a population of healthy females.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female between the ages of 18 and 49 years (at lease 21 subjects) or 50-60 years (no more than 9 subjects);
* Subject is using adequate non-barrier method of birth control [established us of hormonal methods of contraception (oral, injected, implanted, or patch), intrauterine device (IUD) or intrauterine system (IUS), surgical sterilization (e.g. in a monogamous relationship with male partner with vasectomy];
* Subject is free of any vaginal disorders;
* Subject is sexually active and in a monogamous, heterosexual relationship, and whose male partner is willing and able to give informed consent and agrees to engage in sexual intercourse at least twice each week during the two-week study (at least 50% and up to 100% of the study population) or is not sexually active (no more than 50% of the population);
* Subject is a personal lubricant user and agrees to replace her usual personal lubricant with the investigational product;
* Subject has normal menstrual cycle and is not expected to menstruate 2-4 days before or after the examination days;
* Subject agrees to use the provided investigational product at least four times weekly (including at least twice weekly during sexual intercourse for subjects with monogamous, male partners) over the two-week study period;
* Subject exhibits no clinically significant evidence of vulvar or vaginal irritation, as determined by a study doctor, and no reports of sensory irritation at the baseline examination;
* Subject is willing to refrain from introducing any new vaginal products, or using vaginal medication or local contraceptives (including condoms and hormonal rings), during the course of this study;
* Subject agrees to refrain from douching or using any medications, powder, lotions or personal care products in the vulvar or perianal area for the duration of the study (Note: subjects may continue to use their usual pantyliner, if any);
* Subject is willing to use a urine pregnancy test provided to them at baseline and on the third visit (Week 2, day 14);
* Subject has a standard Clinical Research Laboratories, Inc. (CRL) Medical History form on file at CRL and has completed study specific Medical History and Screener/Inclusion forms;
* Subject has signed and, if sexually active and in a monogamous relationship, whose partner has signed, an Informed Consent Form (ICF) in compliance with 21 CFR Part 50: "Protection of Human Subjects";
* Subject (and male partner, if applicable) has completed a HIPAA Authorization Form in conformance with 45 CFR Parts 160 and 164;
* Subject is dependable and able to follow directions as outlined in the protocol;
* Subject receives a score of 0 or 0.5 for erythema and edema, and 0 for sensorial irritation (burning, stinging, itching, and dryness) during the first examination.

Exclusion Criteria:

* Subject is pregnant, nursing, or planning a pregnancy;
* Subject is post-menopausal or has had a hysterectomy;
* Subject is currently using, or has used within two weeks prior to study initiation, any systemic or topical corticosteroids, vasoconstrictors, antibiotics, anti-inflammatories, or antihistamines;
* Subject has known allergies to vaginal or any cosmetic products (including lotions, moisturizer, powder, sprays, etc.);
* Subject reports a history of recurrent bladder, vaginal infection, or incontinence;
* Subject exhibits or reports gynecological abnormalities or has had vaginitis within 60 days prior to study initiation.
* Subject is expected to menstruate 2-4 days before or after the time of the first, second, and third examination;
* Subject uses a vaginal ring, diaphragm or cervical/vault caps, condoms, or condoms with spermicide as a means of contraception;
* Subject has participated in a study involving the vaginal area or in an investigational systemic drug study within two weeks of study initiation;
* Subject receives a score higher than 0.5 for erythema, edema, or >0 for burning, stinging, or itching, during the first examination or shows any other sign of mucosal irregularities (dryness, papules, vesticulation, fissure).

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Laboratories, Piscataway, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Novel Lubricant Miami w/ Frag Personal Lubricant: Healthy subjects use Novel lubricant Miami w/ frag Personal lubricant at least 4 times per week for 2 weeks.
Period: Overall Study
Arm/Group | Novel Lubricant Miami w/ Frag Personal Lubricant
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Novel Lubricant Miami w/ Frag Personal Lubricant
Number analyzed (Participants) | 30
Age, Customized [Number; unit: participants]
  24-59 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Observed Local Erythema
Description: Number of participants with observed erythema by OB/GYN examination.
Time Frame: 14 Days
Population: female only
Measure: Number; unit: participants
Groups:
- Miami w/ Frag Personal Lubricant: Healthy subjects use Miami w/ frag Personal lubricant at least 4 times per week for 2 weeks.
Arm/Group | Miami w/ Frag Personal Lubricant
Number analyzed (Participants) | 30
participants | 0

2. Primary Outcome: Number of Participants With Observed Local Edema
Description: Number of participants with observed edema by OB/GYN examination.
Time Frame: 14 Days
Population: female only
Measure: Number; unit: participants
Arm/Group | Miami w/ Frag Personal Lubricant
Number analyzed (Participants) | 30
participants | 0

ADVERSE EVENTS:
Arm/Group | Miami w/ Frag Personal Lubricant
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Master service agreement and confidentiality agreement in place